CLINICAL TRIAL: NCT07361081
Title: Protocol-Driven Continuous Infusion Versus Intermittent Bolus Heparin During Atrial Fibrillation Ablation
Acronym: AF HEPARIN
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202208043RINB
Record Dates: First submitted 2026-01-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Ablation
Keywords: Atrial Fibrillatio; ablation; Heparin protocol
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thromboembolism and bleeding are still the most common encountered complications during atrial fibrillation ablation. The purpose of this study is to investigate a prespecified protocol-driven continuous heparin infusion method comparing intermittent bolus method for an optimal activated clotting time (ACT) in patients during atrial fibrillation (AF) ablation in Asia population. This is a single-center and retrospective cohort study. The prespecified optimal ACT in this study is defined as 250-350 s. The primary outcome is the frequency of achieving optimal ACT during ablation. Safety outcomes are thromboembolic and major or minor bleeding events during or after ablation. Generalized Estimating Equations (GEE) logistic models will be used to analyze the factors associated with insufficient or over ACT events.

DETAILED DESCRIPTION:
This is a single-center and retrospective cohort study. The study will enroll patients above 20 years old and received RF ablation for AF from 2018 to the end of 2020. The baseline characteristics of the patients will be obtained from the electronic medical records, including age, sex, body weight, body height, risk factors of stroke, cardiac echo, laboratory data, and medications. Three experienced attending physicians are involved in the study. Two used the prespecified continuous infusion protocol to adjust heparin doses.

ELIGIBILITY:
Inclusion Criteria:

1. Above 20 years old
2. Received RF ablation for AF from 2018 to the end of 2020

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center and retrospective cohort study. The study will enroll patients above 20 years old and received RF ablation for AF from 2018 to the end of 2020. The baseline characteristics of the patients will be obtained from the electronic medical records, including age, sex, body weight, body height, risk factors of stroke, cardiac echo, laboratory data, and medications. Three experienced attending physicians are involved in the study. Two used the prespecified continuous infusion protocol to adjust heparin doses.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the frequency of optimal ACT during whole procedure | 400DAYS
  The primary outcome of this study is the frequency of optimal ACT during whole procedure. The prespecified optimal ACT in this study is defined as 250-350s.

SECONDARY OUTCOMES:
Other effective outcomes | 3 days
  total and initial dose of heparin, total heparin and optimal ACT time, average and standard deviation (SD) of ACT, duration of achieving an optimal ACT, and insufficient, optimal and over ACT after loading heparin.
Safety outcomes | 400DAYS
  Manually reviewed by medical records for thromboembolic and major or minor bleeding during or after ablation.
  Any reason delaying hospital discharge would be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital,, Taipei, Taiwan